CLINICAL TRIAL: NCT01537107
Title: Phase I Trial of The Combination of Vismodegib and Sirolimus
Brief Title: Sirolimus and Vismodegib in Treating Patients With Solid Tumors or Pancreatic Cancer That is Metastatic or Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1111; NCI-2011-03809 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-02-14; First posted 2012-02-23 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IV Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — HhAntag691; Sirolimus; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive sirolimus PO QD and vismodegib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vismodegib; Drug: sirolimus; Procedure: positron emission tomography; Procedure: computed tomography; Other: pharmacological study; Other: laboratory biomarker analysis; Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Drug: vismodegib — Given PO
  Other Names: GDC-0449
Drug: sirolimus — Given PO
  Other Names: Rapamune; rapamycin; RAPA
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Correlative studies
  Other Names: tomography, computed
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG

SUMMARY:
This phase I trial studies the side effects and the best dose of sirolimus when given together with vismodegib in treating patients with solid tumors or pancreatic cancer that is metastatic or cannot be removed by surgery. Sirolimus and vismodegib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated dose (MTD) of the combination of vismodegib and sirolimus in unresectable solid tumors. (Cohort I)

SECONDARY OBJECTIVES:

I. To describe the adverse event profile associated with this treatment combination.

II. To describe the tumor responses to treatment combination.

CORRELATIVE OBJECTIVES:

I. To assess the effect of the sirolimus and vismodegib combination on selected biomarkers in tumor biopsies of patients with metastatic pancreatic cancer.

II. To assess the effect of the combination of vismodegib and sirolimus on fludeoxyglucose F 18 (F18-FDG) positron emission tomography (PET) or PET/computed tomography (CT) imaging in Cohort II (MTD) patients with metastatic pancreatic cancer.

III. To study the association of clinical (toxicity and/or tumor response or activity) with the biologic (pharmacodynamic) results obtained by examining tissue biopsies and PET or PET/CT imaging from the same patients.

OUTLINE: This is a dose-escalation study of sirolimus.

Patients receive sirolimus orally (PO) once daily (QD) and vismodegib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* COHORT I (DOSE ESCALATION): histologic proof of cancer that is now unresectable, not amenable to any other standard therapies, or patient refuses standard therapy
* COHORT II (MTD): metastatic adenocarcinoma of the pancreas and tumor amenable to biopsies; prior systemic treatment for metastatic disease is allowed
* Absolute neutrophil count (ANC) => 1500/uL
* Platelet >= 100,000/uL
* Total bilirubin =< upper limit of normal (ULN) Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x ULN
* Creatinine =< 1.5 x ULN
* Hemoglobin >= 9.0 g/dL
* Prothrombin time (PT)/international normalized ratio (INR) < 1.25 x ULN (Cohort II [MTD] only)
* Cholesterol < Common Terminology Criteria for Adverse Events (CTCAE) grade 3
* Triglycerides < CTCAE grade 2
* Magnesium >= lower limit of normal (LLN) and =< ULN
* Ability to provide informed consent
* Willing to return to Mayo Clinic for follow up
* Life expectancy >= 12 weeks
* Cohort II (MTD) only - Translational Research: Willing to provide the biologic specimens as required by the protocol; Note: this is part of the mandatory translational research component
* Women of childbearing potential only: Negative serum pregnancy test done =< 7 days prior to registration; NOTE: female subjects who are pregnant or nursing are excluded from this study; there is no specific mitigation strategy for vismodegib toxicity; however, male patients should be made aware of it during the consent process; although this effect is expected to be reversible with discontinuation of dosing, long-term effects on male fertility cannot be excluded at this time
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Able to swallow or have medication administered through a G-tube and absorb the medication
* Participant agrees to use acceptable form of contraception during the study and for up to 7 months after last study drug dose
* Acceptable forms of contraception:

  * Latex condom (always used with spermicide)
  * Diaphragm (always used with spermicide)
  * Cervical cap (always used with spermicide)
* Acceptable forms of secondary contraception, when used along with a barrier method:

  * Hormonal contraception methods, including pills, patches, rings, or injections except progestin-only containing pills (i.e. "Mini-pill")
  * Tubal ligation
  * Partner's vasectomy
  * Intrauterine device (non-progesterone T)
  * Vaginal sponge (containing spermicide)
* Other acceptable forms:

  * 100% commitment to abstinence
* Unacceptable forms of contraception for women of childbearing potential:

  * Oral contraception containing progestins only
  * Intrauterine device (IUD) progesterone T
  * Female condom
  * Natural family planning (rhythm method) or breastfeeding
  * Fertility awareness
  * Withdrawal
  * Cervical shield
* Willing not to smoke
* Willing to complete a pill diary each day

Exclusion Criteria:

* COHORT I (DOSE ESCALATION): Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes mellitus or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to registration
  * Mitomycin C/nitrosoureas =< 6 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
  * Radiation to > 25% of bone marrow
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Uncontrolled Seizure Disorder
* Central nervous system (CNS) metastases if not stable for at least 2-3 months based on imaging, clinical assessment, use of steroids, or seizure disorder
* Any of the following:

  * Pregnant women
  * Nursing women
  * This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown
* Other concurrent chemotherapy, immunotherapy, radiotherapy, any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) or receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450 3A4 (CPY450 3A4); use of the following strong or moderate inhibitors are prohibited:
* Strong Inhibitors of CYP3A4: Indinavir, Nelfinavir, Ritonavir, Clarithromycin, Itraconazole, Ketoconazole, Nefazodone, Saquinavir, Telithromycin

  * Moderate Inhibitors of CYP3A4: Aprepitant, Erythromycin, Fluconazole, Grapefruit juice, Verapamil, Diltiazem
* Receiving any medications or substances that are inducers of CYP450 3A4

  * Inducers of CYP3A4: Efavirenz, Nevirapine, Carbamazepine, Modafinil, Phenobarbital, Phenytoin, Pioglitazone, Rifabutin, Rifampin, St. John's wort
* Receiving any medications or substances that are strong or moderate inhibitors of CYP450 CYP2C8

  * Strong or Moderate Inhibitors of CYP2C8: Gemfibrozil, Trimethoprim
* Receiving any medications or substances that are inducers of CYP450 2C8

  * Inducer of CYP2C8: Rifampin
* Receiving any medications or substances that are strong or moderate inhibitors of CYP450 CYP2C9

  * Strong or Moderate Inhibitors of CYP2C9: Fluconazole, Amiodarone
* Receiving any medications or substances that are inducers of CYP450 2C9

  * Inducers of CYP2C9: Rifampin, Secobarbital
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients receiving highly active antiretroviral therapy (HAART) treatment
* Active other malignancy, excepting non-melanotic skin cancer or carcinoma-in situ (e.g. of cervix, breast prostate); if there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjogren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Prior therapy with a hedgehog inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
MTD (Cohort I) ) and toxicity profile of combination of vismodegib plus sirolimus every 28 days. | 120 days
  MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients). DLT will be defined as a course 1 adverse event (Common Terminology Criteria for Adverse Events [CTCAE] v 4.0) attributed (definitely, probably, or possibly) to the study treatment. MTD will be examined in an exploratory and hypothesis generating fashion.

SECONDARY OUTCOMES:
Adverse events (AEs) profile in terms of the number and severity of all adverse events (overall, by dose-level, and by tumor group) at baseline, at each dose level and at 30 days after completion of study treatment | 120 days
Time to treatment failure | 120 days
Antitumor effect of molecularly targeted agents non-invasively by F18-FDG PET or PET/CT (Cohort II) | 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Campus in Arizona, Scottsdale, Arizona
  - Mayo Clinic Campus in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota